CLINICAL TRIAL: NCT06610188
Title: The Effect of Inulin on Intestinal Symptoms, Depression and Quality of Life in Individuals With Constipation-Predominant Irritable Bowel Syndrome
Brief Title: The Effect of Inulin in Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mardin Artuklu University (Other)
Responsible Party: Principal Investigator, Çağlar Akçalı, Assist. Prof., Mardin Artuklu University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 377
Record Dates: First submitted 2024-09-19; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Bowel Symptoms; Depression Disorders; Inulin; Constipation; Quality of Life (QOL); Irritable Bowel Syndrome (IBS)
Keywords: Bowel symptoms; depression; inulin; constipation-predominant IBS; quality of life
MeSH Terms: conditions — Constipation; Irritable Bowel Syndrome; Depression | interventions — maltodextrin

STUDY DESIGN:
Intervention Model Description: Individuals were randomly assigned to one of two groups: prebiotic (n=17) and placebo (n=17) groups.
Who Masked: Participant
Masking Description: Participants were blinded to groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prebiotic group (Experimental): products containing a total of 9.2 g (4.6 g twice a day) inulin/oligofructose (50/50) mixture (prebiotic group) that individuals should consume daily were delivered to individuals in identical opaque bags.
  Interventions: Dietary Supplement: Prebiotic group
- Placebo (Placebo Comparator): products containing a total of 9.2 g (4.6 g twice a day) maltodextrin (placebo group) that individuals should consume daily were delivered to individuals in identical opaque bags
  Interventions: Dietary Supplement: Maltodextrin (Placebo)

INTERVENTIONS:
Dietary Supplement: Prebiotic group — products containing a total of 9.2 g (4.6 g twice a day) inulin/oligofructose (50/50) mixture (prebiotic group) that individuals should consume daily were delivered to individuals in identical opaque bags.
  Arms: Prebiotic group
Dietary Supplement: Maltodextrin (Placebo) — products containing a total of 9.2 g (4.6 g twice a day) maltodextrin (placebo group) that individuals should consume daily were delivered to individuals in identical opaque bags.
  Arms: Placebo

SUMMARY:
Purpose: This study was conducted to evaluate the effect of inulin on bowel symptoms, depression and quality of life in individuals with constipation-dominant irritable bowel syndrome. Individuals (n=34) aged 21-63 years with constipation-dominant IBS were included in the study. Individuals were divided into two groups as prebiotic group [(n=17) (inulin/oligofructose 50/50 mixture of 4.6 g (Inulin=total 9.2 g) inulin/oligofructose 50/50 mixture twice a day)], and placebo [(n=17), (Maltodextrin=9.2 g)] group. The intervention period was 8 weeks and Bristol Stool Scale, IBS-Visual Analogue Scale, IBS-Symptom Severity Score Scale (IBS-SSS), IBS-Quality of Life Scale (IBS-QoL) and Beck Depression Scale were administered to the participants at the beginning, 1st month and 2nd month. SPSS software programme was used for statistical analysis of the data. It is thought that inulin supplementation may be effective in reducing symptom severity and frequency, improving bowel function (stool frequency, consistency and transit time) and quality of life, and thus may be beneficial in individuals with constipation-predominant IBS.

DETAILED DESCRIPTION:
In the treatment of IBS, a multimodel perspective that includes psychological support (cognitive behavioural therapy, stress management techniques, etc.) in addition to lifestyle changes (dietary changes, etc.) may be beneficial.

ELIGIBILITY:
Inclusion Criteria:

* the individuals were between 19-65 years of age
* volunteer to participate in the study
* Individuals diagnosed with IBS by a physician according to Rome IV criteria

Exclusion Criteria:

* a history of gastrointestinal surgery (except appendectomy and cholecystectomy)
* inflammatory bowel disease
* lactose malabsorption
* gastroenteritis
* celiac disease
* gastric
* duodenal ulcer
* metabolic diseases (cardiac, hepatic and renal diseases, diabetes, etc.)
* history of malignancy
* pregnancy and lactation
* use of intestinal motility
* antidepressant drugs
* involuntary body weight loss of more than 5 kg in the last 3 months
* use of dietary fibre supplements in the last 3 months
* use of antibiotics in the last 3 months
* use of prebiotic and probiotic supplements in the last 3 months.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
IBS-Visual Analogue Scale (IBS-VAS) | 8 weeks
  The scale, which consists of ten questions in total, is preferred for converting non-numerical values into numerical form. In this scale, the parameter to be evaluated is defined at both ends of a 100 mm line and there are cuts that will enable scoring from 1 to 10. The scoring on the scale indicates that 1:very bad, 10:very good.
The Irritable Bowel Syndrome Symptom Severity Score (IBS/SSS) | 8 weeks
  The Irritable Bowel Syndrome Symptom Severity Score (IBS/SSS) was developed by Francis et al. (1997) to assess the severity of gastrointestinal symptoms in individuals with IBS. It consists of 5 questions in total and each question is scored between 0-100. The IBS-SSS scale has a maximum score of 500 points, which is classed as '75-174 points= mild IBS', '175-299 points= moderate IBS', and '>300 points= severe IBS'.
Irritable Bowel Syndrome Quality of Life Scale (IBS-QoL) | 8 weeks
  The quality of life levels were assessed using the Irritable Bowel Syndrome Quality of Life Scale (IBS-QoL). The Irritable Bowel Syndrome Quality of Life Scale developed by Patrick et al. (1998) is divided into 8 sub-parametres, 34 questions in total and the lowest score is 34, while the highest score is 170. The increase in the total score obtained from the scale indicates a decrease in the quality of life associated with the disease.
The Bristol Stool Scale | 8 weeks
  The Bristol Stool Scale was used to determine the type of IBS through stool forms. This scale aims to predict the stool form over 7 different stool forms. Constipation- predominant IBS was evaluated over the first 4 stool forms, and it is understood that there is an improvement as the stool forms of the individuals approach the type 4 form.
The Beck Depression Scale | 8 weeks
  The Beck Depression Scale was used to evaluate the depression status of the individuals. It is a 21-question (multiple-choice) self-report scale developed by Aaron T. Beck to provide a quantitative assessment of depression severity (Beck, 1961). It provides a four-point Likert-type measurement. The score scale ranges from 0-3 for each question. Total score varies between 0-63. Higher scores obtained from the scale indicate more depressive symptoms. According to the validity and reliability article of the scale for Turkish, it was stated that the cut-off score was accepted as 17. In this study, the data were divided into two groups as depressed and non-depressed according to the scale using a cut-off score of 17.

CONTACTS AND LOCATIONS:
Locations (1):
- Mardin Artuklu University, Mardin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data will not be shared because it contains personal information.